CLINICAL TRIAL: NCT05572697
Title: App-delivered Cognitive-behavioral Therapy for Insomnia Among Patients With Comorbid Musculoskeletal Complaints and Insomnia Referred to 4-week Inpatient Multimodal Rehabilitation
Brief Title: App-delivered Cognitive-behavioral Therapy for Insomnia Among Patients With Musculoskeletal Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 496297
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Insomnia; Pain, Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Cluster randomized clinical trial with two parallel arms
Masking Description: Outcomes will be measured by registry data and questionnaires. Researchers will not have access to the randomization key before analyses are performed but blinding is not possible due to different number of participants in the two groups (as randomization is 2:1). The randomization procedure will be performed by the Clinical Research Unit (Klinforsk) at The Faculty of Medicine and Health Sciences at the Norwegian University of Science and Technology (NTNU) by use of a computer-generated block randomization. The randomization will be on group level to avoid contamination between participants in the same rehabilitation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Cognitive-behavioral therapy for insomnia (dCBT-I) (Experimental): In addition to the standard rehabilitation program, participants will receive the sleep intervention delivered via a smartphone app. We will use a Norwegian a program named Assistert Selvhjelp (In English: "Assisted Self-Help"). The app is fully automated and requires no contact with healthcare personnel. It can also be assessed on computers, but in the present project we will use the app-delivered version. It is based on the principles from face-to-face CBT-I including several modules consisting of sleep hygiene, stimulus control sleep restriction, cognitive therapy, and relaxation training. The modules also consist of learning material (e.g., quizzes and materials explaining and educating the patients about important sleep dimensions).
  Interventions: Behavioral: Digital Cognitive-behavioral therapy for insomnia (dCBT-I)
- Usual care (Active Comparator): Participants randomized to usual care will receive the standard inpatient rehabilitation program. This is a traditional rehabilitation program consisting of physical activity, mindfulness excises, psychoeducation and acceptance and commitment therapy. One of the educational sessions is about sleep. Although this educational session overlaps with some of the content included in the intervention (e.g., sleep hygiene, stimulus control), it does not include any of the interactive features of the app.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Digital Cognitive-behavioral therapy for insomnia (dCBT-I) — 6 week sleep intervention delivered via a smartphone app while taking part in inpatient multimodal rehabilitation for chronic pain lasting 2+2 weeks.
  Arms: Digital Cognitive-behavioral therapy for insomnia (dCBT-I)
Behavioral: Usual care — Inpatient multimodal rehabilitation for chronic pain lasting 2+2 weeks.
  Arms: Usual care

SUMMARY:
The aim of this randomized clinical trial is to evaluate the effectiveness of app-delivered cognitive-behavioral therapy for insomnia adjunct to inpatient multimodal rehabilitation for individuals with comorbid insomnia and chronic pain, compared with rehabilitation (usual care) only.

DETAILED DESCRIPTION:
Insomnia is highly prevalent among patients receiving treatment for long-term musculoskeletal complains. Cognitive-behavioral therapy for insomnia (CBT-I) may be effective for improving sleep quality and pain-related outcomes in these patients, but the availability of this therapy is limited by few trained therapists. In this randomized clinical trial we will evaluate the effectiveness of app-delivered CBT-I adjunct to inpatients multimodal rehabilitation for individuals with comorbid insomnia and chronic pain, compared with rehabilitation (usual care) only. Patients referred to Unicare Helsefort (Norway) with long-term chronic musculoskeletal complains and insomnia are invited to the study. The rehabilitation program consists of 2+2 weeks of inpatient multimodal rehabilitation, where the patients are at home for two weeks between the rehabilitation stays. Participants in the intervention group will receive the (CBT-I) while participating in rehabilitation, while the control group will receive rehabilitation without the app (usual care).

Based on sample size calculation recruiting 15 clusters with 2:1 randomization will achieve 80 % power to detect a 4-point difference between the intervention and usual treatment group on the insomnia severity index (ISI).

Edit 25.08.23: We noted in the review process of a protocol paper that the description of our sample size calculation implied that 150 participants would be included in the study, rather than that 150 potential participants would be screened and that we anticipated that 5 from each group of the 15 clusters would be eligible (i.e. 75 included in the study). We have also revisited the sample size calculations to account for dropouts and low adherence rates known to be a problem in digital interventions. We expect a dropout rate of approximately 20 % and that around 50 % of the participants in the intervention group will complete at least four of the dCBT-I modules. Given that the per-protocol analysis is of particular interest in this study, we aim to recruit 21 clusters to account for the fact that we expect an average of four participants per cluster in the control group to complete the follow-up, and an average of two participants in the intervention group to complete at least four of the modules and attend the follow-up. As total sample size is hard to predict and the sample size is based on number of clusters we have not changed the total enrollment number.

ELIGIBILITY:
Inclusion Criteria:

* Taking part in inpatient rehabilitation due to long-term musculoskeletal complaints
* Insomnia Severity Index (ISI) score >11.

Exclusion Criteria:

* Not having a smartphone or tablet.
* Individuals with work schedules that includes night shifts during the intervention
* Pregnancy
* Inadequate opportunity to sleep or living circumstances that prevent modification of sleep patterns such as having an infant
* Currently receiving psychological treatment for insomnia
* Medical history of contraindicating use of CBT-I such as epilepsy, recent cardiac surgery, and an attack phase of multiple sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Insomnia | 3 months of follow-up
  Degree of sleep problems measured by the insomnia severity index (ISI).

SECONDARY OUTCOMES:
Insomnia | Measured at 3, 6 and 12 months of follow-up, main assessment at 3 months
  Difference in the proportion of participants that achieves an 8-point improvement in their Insomnia Severity Index -score between inpatient multidisciplinary rehabilitation + dCBT-I (intervention group) and inpatient multidisciplinary rehabilitation only (control group).
Insomnia | 6 and 12 months of follow-up
  Degree of sleep problems measured by the insomnia severity index (ISI).
Health-related quality of life | 3, 6 and 12 months of follow-up, main assessment at 3 months
  Measured by the EuroQol EQ5D-5L questionnaire
Pain intensity | 3, 6 and 12 months of follow-up, main assessment at 3 months
  Scored from 0-100 on a visual analogue scale
Sick leave | 12 months of follow-up
  Registry data from the National Insurance Administration (NAV).
Use of sleep and pain medications | 12 months of follow-up
  Data from the national prescription registry
Physical function | 3, 6 and 12 months of follow-up, main assessment at 3 months
  Measured by the Patient-Specific Functional Scale (PSFS). Scored 0-10.
Fatigue | 3, 6 and 12 months of follow-up, main assessment at 3 months
  Scored from 0-100 on a visual analogue scale
Physical activity | Measured at 3, 6 and 12 months of follow-up, main assessment at 3 months
  Physical activity measured by a questionnaire adapted from the Trøndelag Health Study (HUNT Study) which consists of three questions about frequency, duration and intensity of physical activity per week.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Aasdahl, Principal Investigator — Norwegian University of Science and Technology; Solveig K Grudt, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Unicare Helsefort, Rissa, Hasselvika, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skarpsno ES, Simpson MR, Seim A, Hrozanova M, Bakoy MA, Klevanger NE, Aasdahl L. App-Delivered Cognitive-Behavioral Therapy for Insomnia Among Patients with Comorbid Musculoskeletal Complaints and Insomnia Referred to 4-Week Inpatient Multimodal Rehabilitation: Protocol for a Randomized Clinical Trial. Nat Sci Sleep. 2023 Oct 11;15:799-809. doi: 10.2147/NSS.S419520. eCollection 2023. PMID 37850197

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT05572697/SAP_001.pdf